CLINICAL TRIAL: NCT05408442
Title: Role of Pulmonary Perfusion on Tolerance to Supine Position in Patients With Acute Respiratory Distress Syndrome on Mechanical Ventilation
Brief Title: Role of Pulmonary Perfusion on Tolerance to Supine Position in Patients With ARDS
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Maria Consuelo Bachmann, Principal investigator, Pontificia Universidad Catolica de Chile
Other Study IDs: 210309002
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: ARDS; Mechanical Ventilation; Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prone: ARDS patients during mechanical ventilation in prone position
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The relationship between the presence or absence of endothelial dysfunction and changes in pulmonary perfusion will be evaluated, to then determine if there is any association between changes in the V / Q ratio and tolerance to the supine position after a prone cycle in patients with acute respiratory distress syndrome on mechanical ventilation.

DETAILED DESCRIPTION:
The prone position is a strategy used in patients with respiratory failure in order to improve oxygenation, it has proven to be very effective compared to the supine position, reducing mortality in critically ill patients diagnosed with acute respiratory distress syndrome. Physiologically, these clinical findings could be explained by an improvement in the ventilation/perfusion ratio (V/Q). Animal studies have shown that the prone position significantly decreases the collapse of the dorsal regions of the lung, the one that anatomically receives the highest percentage of blood flow. Nevertheless, to this day the physiology behind these benefits in critically ill patients has not been studied, and without this, the indications for use or duration of the maneuver has not yet been determined.

For many intensivists, determining the best time to re-supinate the patient is one of the greatest challenges they face in clinical practice, since intolerance to supine position and the need for a new prone cycle has been associated to the risk of complications, such as accidental extubation, hemodynamic instability and intensive care unit (ICU) acquired weakness. For this reason, it is relevant to determine what factors are associated with tolerance to supine position, and knowing the presence of vascular defects due to endothelial dysfunction during conventional and COVID-19 ARDS, our hypothesis is that patients who do not tolerate the change to supine position after a prone cycle are unable to maintain an optimal V/Q ratio, this due to the loss of regulation of the hypoxic pulmonary vasoconstriction phenomenon related to endothelial dysfunction markers.

For this observational cohort clinical study, patients admitted to the intensive care unit of the UC-CHRISTUS Clinical Hospital with diagnosis of ARDS will be evaluated. After inclusion and the signing of the informed consent, physiological data of the patients will be recorded. In addition, an evaluation of vascular function will be performed through ultrasound, near infrared spectroscopy, and markers of endothelial damage in plasma. After baseline measurements, the distribution of pulmonary ventilation and perfusion through EIT, pulmonary function, hemodynamic, ventilatory and arterial gases will be evaluated. These measurements will be taken again 1 hour before to position change, and 1, 8, 12 and 24 hours after the change to supine position.

With this study the investigators hope to be able to find a pattern associated to endothelial function and perfusion in these patients that allows us to determine which patient can be repositioned supine, without the need for a new prone cycle. With this information, an evaluation and management protocol could be developed at long term for patients subjected to prone position, which allows less time in mechanical ventilation and a reduction of the complications and risks associated with the maneuver and with the ICU length of stay that directly affects the quality of life of these patients in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ARDS
* Patients connected to IMV
* Patients in prone position for less than 48 hours.

Exclusion Criteria:

* Diagnosis of exacerbation of chronic lung disease or cardiogenic pulmonary edema.
* Presence of contraindications for the use of the prone position and for the use of the EIT belt
* Patient under 18 years of age
* Pregnancy
* Refusal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the ICU of Hospital Clínico Universidad Católica
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Tolerance to supine position | 12 hours
  It will be defined by changes in PaO2/FiO2 after position changes

SECONDARY OUTCOMES:
Endothelial dysfunction | 48 hours
  Presence of endothelial dysfunction markers in plasma (angiopoietin-1)
V/Q changes | 48 hours
  Changes in ventilation/perfusion ratio
Endothelial dysfunction | 48 hours
  Presence of P-selectin in plasma
Endothelial dysfunction | 48 hours
  Presence of E-selectin in plasma
Endothelial dysfunction | 48 hours
  Presence of VCAM-1 in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad Católica, Santiago, Santiago Metropolitan, Chile